CLINICAL TRIAL: NCT06313229
Title: Simultaneous Versus Staged Implant Placement With Vertical and Horizontal Bone Augmentation Using Autogenous Cortical Bone Plates Combined With a Mixture of Platelet-rich Fibrin and Allobone Grafts.
Brief Title: Simultaneous Implant Placement With Vertical and Horizontal Bone Augmentation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-195
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Bone Loss; Dental Implant Failed
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: single-center, prospective, single-blinded, randomized parallel two-arm controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The present clinical trial was single-blinded one as the evaluator and the statistician were both blinded. While both the implantologist or the participant were not blinded as the interventions were dissimilar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staged implant placement approach (Experimental): the bone defect was grafted using bone plates buccally and palatally and the defect between plates was grafted by sticky allogenic bone graft. 6 months later the implant was placed in the grafted site.
  Interventions: Procedure: implant placement 6 months after ridge augmentation
- Simultaneous implant placement approach (Experimental): the bone defect was grafted using bone plates buccally and palatally and the defect between plates was grafted by sticky allogenic bone graft combined with simultaneous implant placement.
  Interventions: Procedure: implant placement Simultaneously with ridge augmentation

INTERVENTIONS:
Procedure: implant placement 6 months after ridge augmentation — the deficient ridge was grafted first followed by implant placement after 6-monthes
  Arms: Staged implant placement approach
Procedure: implant placement Simultaneously with ridge augmentation — the deficient ridge was grafted and followed by implant placement simultaneously
  Arms: Simultaneous implant placement approach

SUMMARY:
The purpose of this study was to report the clinical and radiographical outcomes of using autogenous cortical bone plates combined with sticky allogenic bone graft for augmenting maxillary anterior atrophic combined horizontal and vertical ridge defects with simultaneous versus staged implant placement.

DETAILED DESCRIPTION:
Sufficient alveolar ridge is a prerequisite for successful implant stability, atrophic ridges defects make the placement of regular implants challenging. A variety of materials and surgical techniques are available for bone augmentation procedures prior implant placement. The present study evaluated the effect of sticky allogenic bone graft for the horizontal and vertical ridge augmentation with simultaneous implant placement using autogenous cortical bone plates in maxillary anterior atrophic ridge defects.

Forty-two patients, with severe maxillary anterior horizontal and vertical atrophic ridge deficiencies were randomly assigned to two groups: staged approach group and simultaneous implant placement group. The two groups were grafted using bone plated buccally and palatally and the defect between plates was grafted by sticky allogenic bone graft. Radiographic examination was performed immediately before bone grafting procedure and at 6, 12 months postoperatively, to evaluate the change of bone width and height.

ELIGIBILITY:
Inclusion Criteria:

* Good general health at the time of surgery
* At least 3 months of healing after tooth extraction
* Horizontally and vertical compromised alveolar ridges

Exclusion Criteria:

* Thick cortex in the labial/buccal with less cancellous bone inside;
* Obvious undercut on the labial/buccal side
* Uncontrolled periodontal conditions or other oral disorders;
* history of radiotherapy in the head and neck region

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
Stability Quotient of Implants (SQI) | 12-month.
  The implant stability was recorded using Osstell TM. Following implant insertion, SQI readings were taken immediately, then again after six and twelve months.
Horizontal bone dimensions (HBDs) | 12-month.
  The HBD alterations were assessed by measuring horizontal spacing between the external edges of labial and palatal bony plates at a level 2mm apical of the fixture platform.
Peri-implant Bone Density (PBD) | 12-month.
  For consistent measurement of the PBD, 1-mm-diameter Region of interest (RI) was selected and traced 1.2 mm distant from the fixture on the cross-sectional slices followed by counting the threshold pixels inside the RI.

CONTACTS AND LOCATIONS:
Overall Officials: Walid AH Elamrousy, PhD, Principal Investigator — Faculty of Oral and Dental Medicine, Kafrelsheikh University
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided